CLINICAL TRIAL: NCT01270750
Title: Pilot Trial of Bosentan for Secondary Pulmonary Hypertension Due to Severe Mitral Valve Dysfunction
Brief Title: Bosentan for Severe Mitral Valve Dysfunction
Acronym: BOSMIVAR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Chalkida (Other Government)
Responsible Party: GEORGE VLACHOGIORGOS, General Hospital of Chalkida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHC2/29/22-09-2008
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: SECONDARY PULMONARY HYPERTENSION; MITRAL STENOSIS; CHILDHOOD RHEUMATOID FEVER; CONGESTIVE HEART FAILURE
Keywords: ENDOTHELIN RECEPTOR ANTAGONIST; BOSENTAN; SECONDARY PULMONARY HYPERTENSION; RHEUMATOID FEVER; CONGESTIVE HEART FAILURE; SECONDARY PULMONARY HYPERTENSION DUE TO MITRAL STENOSIS
MeSH Terms: conditions — Mitral Valve Stenosis; Heart Failure | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BOSENTAN — TWICE DAILY PERORAL BOSENTAN, 125 MG DAILY DIVIDED IN TWO DOSES DURING THE FIRST MONTH AND 250 MG DAILY DIVIDED IN TWO DOSES SUBSEQUENTLY.

SUMMARY:
Vasoconstrictive signaling via endothelin receptors is not limited to primary pulmonary arterial hypertension, but has also been documented in secondary pulmonary hypertension due to congestive heart failure, including cardiac valve disease. The investigators aim to examine the clinical and physiologic effects of bosentan therapy in patients with secondary pulmonary hypertension due to severe, inoperable cardiac valve disease, using a single-center, prospective, open-label, non-randomized study of oral bosentan in outpatients with severe mitral stenosis due to childhood rheumatoid fever. Primary end-point will be exercise capacity at six months determined by six-minute walking distance and cardiopulmonary exercise testing. Secondary end-points will be symptomatic relief, echocardiographic left ventricular function and pulmonary pressure, serum pro-brain natriuretic peptide, and adverse events at six months.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* > 60 Yrs Old
* < 85 Yrs Old
* Stable disease
* Congestive heart failure NYHA IIIB/V
* Inoperable mitral stenosis due to childhood rheumatoid fever
* Mean pulmonary artery pressure > 40 cm H2O

Exclusion Criteria:

* Prior treatment with endothelin receptor antagonist(s)
* Hospitalization (exacerbation)
* Cardiac valve surgery

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
SIX MINUTE WALKING DISTANCE | SIX MONTHS
  CHANGE IN SIX MINUTE WALKING DISTANCE AFTER 6 MONTHS OF THERAPY COMPARED TO PRE-TREATMENT VALUE.
MAXIMAL OXYGEN UPTAKE | 6 MONTHS
  CHANGE IN MAXIMAL OXYGEN UPTAKE AFTER 6 MONTHS OF THERAPY COMPARED TO PRE-TREATMENT VALUE.

SECONDARY OUTCOMES:
ECHOCARDIOGRAPHIC PULMONARY PRESSURE | 6 MONTHS
  ECHOCARDIOGRAPHIC ASSESSMENT OF PEAK AND MEAN PULMONARY PRESSURE AT 6 MONTHS AFTER TREATMENT COMPARED WITH PRE-TREATMENT VALUES.
ECHOCARDIOGRAPHIC LEFT VENTRICULAR FUNCTION | 6 MONTHS
  ECHOCARDIOGRAPHIC ASSESSMENT OF LEFT VENTRICULAR FUNCTION AT 6 MONTHS AFTER TREATMENT COMPARED WITH PRE-TREATMENT VALUES.
SERUM PRO-BNP | 6 MONTHS
  ASSESSMENT OF SERUM PRO-BRAIN NATRIURETIC PEPTIDE LEVELS AT 6 MONTHS AFTER TREATMENT COMPARED WITH PRE-TREATMENT VALUES.
DYSPNEA | 6 MONTHS
  CHANGE IN BORG DYSPNEA INDEX COMPARED WITH PRE-TREATMENT VALUES.

CONTACTS AND LOCATIONS:
Overall Officials: GEORGE VLACHOGIORGOS, MD PHD, Principal Investigator — GENERAL HOSPITAL OF CHALKIDA, GREECE
Locations (1):
- General Hospital of Chalkida, Chalcis, Evoia, Greece